CLINICAL TRIAL: NCT04312672
Title: Long-term Follow-up Study of Participants Following an Open Label, Multi-Centre, Phase I/II Dose Escalation Trial of a Recombinant Adeno-associated Virus Vector (AAV5- hRKp.RPGR) for Gene Therapy of Adults and Children With X-linked Retinitis Pigmentosa Owing to Defects in Retinitis Pigmentosa GTPase Regulator (RPGR)
Brief Title: Long-term Follow-up Gene Therapy Study for RPGR- XLRP
Status: Completed | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: MGT010; MGT010 (Other: Janssen Research & Development, LLC); 2018-000425-31 (EudraCT Number)
Record Dates: First submitted 2019-07-15; First posted 2020-03-18 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: X-Linked Retinitis Pigmentosa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Follow up cohort: no intervention follow up study
  Interventions: Biological: AAV5-hRKp.RPGR

INTERVENTIONS:
Biological: AAV5-hRKp.RPGR — Participants will not receive any intervention in this study. Participants from the retrospective (MGT009-NCT03252847) study will be follow-up.

SUMMARY:
This is a long-term follow-up study assessing safety of patients for up to 60 months following advanced therapy investigational medicinal product (ATIMP) AAV5-hRKp.RPGR vector in participants with XLRP caused by mutations in RPGR.

ELIGIBILITY:
Inclusion Criteria:

* Received AAV5-hRKp.RPGR in the MGT009 Study

Exclusion Criteria:

* Unwilling or unable to meet with the requirements of the study

Min Age: 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Males receiving AAV5-hRKp.RPGR in the MGT009 study
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2025-09-17 (Actual); Study Completion 2025-09-17 (Actual)

PRIMARY OUTCOMES:
Assess the Longer-term Safety of AAV5-hRKp.RPGR Administered to Participants | 60 Months
  Longer-term safety of subretinal AAV5-hRKp.RPGR administered to participants will be reported.

SECONDARY OUTCOMES:
Change in Functional Vision of Walk Time in Vision-guided Mobility Assessment (VMA) | Up to 60 Months
  Change in functional vision of walk time after treatment administration in VMA (Version 1.0) will be reported.
Change in Functional Vision of Low Luminance Questionnaire (LLQ) Domain Scores in Patient Reported Outcome (PRO) | Up to 60 Months
  Change in functional vision of LLQ domain scores in PRO will be reported. The instrument is scored by domain, computed by scaling individual items from 0 to 100 and then averaging the individual items for each domain. A higher score reflects higher functional level.
Change in Best Corrected Visual Acuity (BCVA) Using the Early Treatment Diabetic Retinopathy Study (ETDRS) Chart Letter Score | Up to 60 Months
  The longer-term efficacy of AAV5-hRKp.RPGR in change in BCVA using ETDRS chart letter score will be reported.
Change in Low Luminance Visual Acuity (LLVA) as Assessed by ETDRS Chart Under Low Luminance Conditions | Up to 60 Months
  Change in LLVA as assessed by ETDRS chart under low luminance conditions will be reported.
Change in Mean Retinal Sensitivity Within the Central 10 Degree Visual Field Excluding Scotoma (MRS10) in Static Perimetry | Up to 60 months
  Change in mean retinal sensitivity within the central 10 degrees excluding scotoma (MRS10) in static perimetry will be reported.
Change In Retinal Sensitivity by Pointwise Comparison of Data in Static Perimetry Within the Full Visual Field | Up to 60 months
  Change in retinal sensitivity by pointwise comparison of data in static perimetry within the full visual field will be reported.
Change In Retinal Sensitivity by Pointwise Comparison of Data in Static Perimetry Within the Central 30 Degrees Visual Field | Up to 60 months
  Change in retinal sensitivity by pointwise comparison of data in static perimetry within the Central 30 Degrees visual field will be reported.
Change in Mean Retinal Sensitivity Within the Full Visual Field Excluding Scotoma (MRS90) in Static Perimetry | Up to 60 months
  Change in mean retinal sensitivity within the full visual field excluding scotoma (MRS90) in static perimetry will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (5):
- United States (3):
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - Univ of Michigan Medical Center, Ann Arbor, Michigan
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
- United Kingdom (2):
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Moorfields Eye Hospital, London